CLINICAL TRIAL: NCT01710943
Title: Web-based CBT for Substance Misusing and PTSD Symptomatic OEF/OIF Veterans
Brief Title: Web-based CBT for Recent Veterans Experiencing Problems With Trauma Symptoms or Alcohol/Drug Use
Acronym: Web CBT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: The VA Western New York Healthcare System (U.S. Federal Agency); Syracuse VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrew Rosenblum, Director, Institute for Treatment and Services Research, National Development and Research Institutes, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AA020181 (NIH)
Record Dates: First submitted 2012-04-26; First posted 2012-10-19 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Post-Traumatic Stress Symptoms; Problematic Use of Alcohol or Other Drugs
Keywords: Web-based CBT; PTSD; Alcohol Misuse; Substance Misuse; Integrated Primary Care; OEF/OIF Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based Cognitive Behavioral Treatment (Experimental): Participants who are randomly assigned to the treatment condition will receive the same standard care as those in the control condition and they will also receive access to the web-based CBT intervention. Participants in this condition will be asked to complete 24 CBT sessions, 2 sessions/topics per week for 12 weeks. Participants will be asked to complete the 18 "core modules" of the program during the first 9 weeks of the trial and then to re-visit important modules and complete optional modules of their choice during the final 3 weeks of the trial.
  Interventions: Behavioral: Web-based Cognitive Behavioral Treatment
- Treatment as Usual (No Intervention): TAU consists of the usual Veterans Integrated Service Network 2 (VISN) primary care services. As we have described, all of the participants will be recruited from patients presenting for treatment typically for physical complaints in primary care clinics in VA's VISN 2 (Upstate NY). VISN 2 officially practices a co-located, collaborative care model of integrated (behavioral health and physical health) in its primary care clinics. This integrated model has been implemented widely in both VA and non-VA primary care clinics in the United States .

INTERVENTIONS:
Behavioral: Web-based Cognitive Behavioral Treatment — Participants in this condition will be asked to complete 24 CBT sessions, 2 sessions/topics per week for 12 weeks. We expect that each session will be approximately 30 minutes in duration. Participants will be asked to complete the 18 "core modules" of the program during the first 9 weeks of the trial and then to re-visit important modules and complete optional modules of their choice during the final 3 weeks of the trial. They can choose to do this using a designated computer in a private room at their local VA or can complete these sessions in the privacy of their own home with their personally-owned computers. Participants can choose to complete each session on any day/time of their choosing in a given week.
  Other Names: Web-based CBT
  Arms: Web-based Cognitive Behavioral Treatment

SUMMARY:
The proposed study involves developing and evaluating an interactive, web-based CBT intervention for OEF/OIF Veterans with hazardous or problematic substance use and PTSD symptoms (PTSD or subsyndromal PTSD). The intervention will address the special culture and experiences of the investigators targeted population (OEF/OIF Veterans). The web-based CBT intervention includes 24 modules, to be used across 24 sessions targeting OEF/OIF Veterans with hazardous or problematic substance use and PTSD symptoms. The investigators ask participants to complete 2 sessions per week (one module per session) for 12 weeks. The first 18 modules to be completed across 18 sessions (9 weeks) are considered core modules relevant to all Veterans in the target population. These modules are designed to reduce posttraumatic stress symptoms as well as reduce and prevent the escalation of problematic substance use. The remaining 6 module topics are considered "optional" and are used based on the interest and clinical need of various sub-groups of VA patients. The study includes initial input as well as feedback on a beta version from experts who have worked with OEF/OIF veterans with PTSD and substance abuse problems as well as input/feedback from the target population (the Veterans themselves). In addition to presenting content grounded in evidence-based CBT interventions, the program also employs state of the art technologies to deliver module content grounded in evidence-based learning principles, including Computer-Assisted Instruction, Computer Simulation and other interactive exercises.

ELIGIBILITY:
Phase 1: Focus Groups

Inclusion Criteria:

1. At least 18 years of age
2. An OEF or OIF veteran (verified via CPRS)
3. Screen positive on the Audit-C (>=3 for women or >= 4 for men) OR screen positive on the PC-PTSD (>=3).
4. Currently receiving primary medical care at a VA Medical Center (verified via CPRS)

Exclusion Criteria:

1. Insufficient ability to understand or provide informed consent
2. Lack sufficient ability to use English to participate in the consent process,
3. Current plan or intent to harm themselves as measured with the suicide assessment in Appendix D after the consent process.

Phase 2: Feedback Sessions

Inclusion Criteria

1. At least 18 years of age
2. An OEF or OIF veteran (verified via CPRS)
3. Hazardous or harmful substance use as measured by one of the following:

   * AUDIT-C score of >=3 (for women) or >= 4 (for men) OR
   * DAST score of >=2 OR
   * Have exited a controlled environment (e.g., detoxification unit, hospital, or correctional facility) within 30 days of screening AND within 30 days prior to entering the controlled environment report:

     i. heavy drinking (>3 drinks for women or > 4 drinks for men on one or more days), or ii.use of any illegal drugs, iii.or misuse of prescription drugs (use in excess of the directions or any non-medical use)
4. Screen positive on the PC-PTSD (>=2).
5. Currently receiving primary medical care at a VA Medical Center (verified via CPRS)

Exclusion Criteria:

1. Insufficient ability to understand or provide informed consent
2. Lack sufficient ability to use English to participate in the consent process, the computerized intervention or the assessments.
3. Current plan or intent to harm themselves as measured with the suicide assessment in Appendix D administered after the consent process.

Phase 3: Randomized Clinical Trial

Inclusion Criteria:

1. At least 18 years of age
2. An OEF or OIF veteran (verified via CPRS)
3. Hazardous or harmful substance use as measured by one of the following:

   * AUDIT score of >=7 (for women) or >= 8 (for men) OR
   * DAST score of >=2 OR
   * Have exited a controlled environment (e.g., detoxification unit, hospital, or correctional facility) within 30 days of screening AND within 30 days prior to entering the controlled environment report:

     i. heavy drinking (>3 drinks for women or > 4 drinks for men on1 or more days) or ii. use of any illegal drugs iii. misuse of prescription drugs (use in excess of the directions or any non-medical use)
4. Determined to have diagnostic-level or PTSD (1 A symptom, 1 B symptom, 3 C symptoms AND 2 D symptoms) or subthreshold PTSD (1 A symptom, 1 B symptom, 3 C symptoms OR 2 D symptoms) on the Clinician Administered PTSD Scale (CAPS).
5. Currently receiving primary medical care at a VA Medical Center (verified via CPRS)

Exclusion Criteria:

1. Plans to move out of area within the next three months
2. Currently enrolled in a substance abuse treatment program or receiving treatment for PTSD from a mental health professional (verified via CPRS).
3. Insufficient ability to understand or provide informed consent
4. Lack sufficient ability to use English to participate in the consent process, the computerized intervention or the assessments.
5. In need of alcohol detoxification as determined by a score of > 15 on the Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar).
6. Current plan or intent to harm themselves as measured with the suicide assessment in Appendix D administered after the consent process.
7. Medical chart diagnosis of a current psychotic disorder, including schizophrenia or bi-polar disorder
8. Cognitive impairment specified by a medical chart diagnosis. Diagnoses include dementia and moderate to severe traumatic brain injury (TBI). Patients with mild TBI will not be excluded. The Second Level TBI Assessment present in patient medical records can be used to verify the severity of TBI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptomatology | 12 weeks
  Comparing baseline score of the PCL-M to 12 weeks score
PTSD Symptomatology | 1 month post-intervention
  Comparing baseline score of the PCL-M to score 1 month post-intervention discharge
PTSD Symptomatology | 3 months post-intervention
  Comparing baseline score of the PCL-M to score 3 months post-intervention
Alcohol and Drug Use | 12 weeks
  Comparing baseline score of the Timeline Follow-back (TLFB)to 12 weeks score
Alcohol and Drug Use | 1 month post-intervention
  Comparing baseline TLFB score to score 1 month post-intervention
Alcohol and Drug Use | 3 month post-intervention
  Comparing baseline TLFB score to score 3 month post-intervention
Quality of Life | 12 weeks
  Comparing baseline EuroQOl and WHOQOL-Bref scores to scores at 12 weeks
Quality of Life | 1 month post-intervention
  Comparing baseline EuroQOl and WHOQOL-Bref scores to scores at 1 month post-intervention
Quality of Life | 3 month post-intervention
  Comparing baseline EuroQOl and WHOQOL-Bref scores to scores at 3 months post-intervention
Cost-Effectiveness | 12 weeks
  Cost-effectiveness of web-based intervention compared to standard care, as measured by the Brief DATCAP, EuroQol EQ5D, and Non-Study Medical and Other Services (NSMS) scales

SECONDARY OUTCOMES:
Resiliency and Positive Affect | 12 weeks
  Comparing baseline Connor-Davidson Resilience Scale (CD-RISC) and the Positive Affect Negative Affect Scale (PANAS)scores to scores at 12 weeks
Resiliency and Positive Affect | 1 month post-intervention
  Comparing baseline Connor-Davidson Resilience Scale (CD-RISC) and the Positive Affect Negative Affect Scale (PANAS)scores to scores at 1 month post-intervention
Resiliency and Positive Affect | 3 months post-intervention
  Comparing baseline Connor-Davidson Resilience Scale (CD-RISC) and the Positive Affect Negative Affect Scale (PANAS)scores to scores at 3 months post-intervention
Insomnia | 12 weeks
  Comparing baseline Insomnia Severity Index (ISI)score to score at 12 weeks
Insomnia | 1 month post-intervention
  Comparing baseline score on the Insomnia Severity Index (ISI) to score at 1 month post-intervention
Insomnia | 3 months post-intervention
  Comparing baseline score on the Insomnia Severity Index (ISI) to score at 3 month post-intervention
Psychological Distress | 12 weeks
  Comparing baseline score on the 10-item version of Symptom Checklist-90 (SCL-90) to score at 12 weeks
Psychological Distress | 1 month post-intervention
  Comparing baseline score on the 10-item version of Symptom Checklist-90 (SCL-90) to score at 1 month post-intervention
Psychological Distress | 3 months post-intervention
  Comparing baseline score on the 10-item version of Symptom Checklist-90 (SCL-90) to score at 3 months post-intervention
Pain Severity and Pain Interference | 12 weeks
  Comparing baseline score on the Brief Pain Inventory (BPI) to score at 12 weeks
Pain Severity and Pain Interference | 1 month post-intervention
  Comparing baseline score on the Brief Pain Inventory (BPI) to score at 1 month post-intervention
Pain Severity and Pain Interference | 3 months post-intervention
  Comparing baseline score on the Brief Pain Inventory (BPI) to score at 3 months post-intervention
Treatment Satisfaction | 12 weeks
  As measured using visual analog scales assessing participant's impressions of how useful, interesting, etc. their treatment has been.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rosenblum, Ph.D., Principal Investigator — National Development and Research Institutes, Inc.; Stephen Maisto, Ph.D., Principal Investigator — Syracuse University
Locations (2):
- United States (2):
  - Buffalo VA Medical Center, Buffalo, New York
  - Syracuse VA Medical Center, Syracuse, New York